CLINICAL TRIAL: NCT04223986
Title: Prehospital Risk Stratification in Acute Coronary Syndromes- Feasibility Trial
Brief Title: Prehospital Risk Stratification in Acute Coronary Syndromes
Acronym: Pre-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/05178-2 - 522
Record Dates: First submitted 2018-10-23; First posted 2020-01-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2018-11

CONDITIONS: Acute Coronary Syndrome; Non-ST Elevation Myocardial Infarction (nSTEMI)
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Prospective enrollment on inclusion criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound and Troponin T (Other): 5 images transferred to cardiologist
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: Troponin- T quick test

INTERVENTIONS:
Diagnostic Test: Ultrasound — decide between the need for intervention or not (Percutaneous coronary intervention)
Diagnostic Test: Troponin- T quick test — Quick test for Troponin T blood assessment
  Other Names: Cobas

SUMMARY:
A feasibility study of prehospital echocardiographic examination and point-of-care troponin analysis, conducted by paramedics, in patients with suspected acute coronary syndrome. Echocardiographic images are sent together with information of TnT values and ECG signs to there cardiologist on call, deciding for immediate Cath lab (PCI) evaluation or local hospital evaluation.

DETAILED DESCRIPTION:
Assessing the feasibility and sensitivity and specificity of prehospital risk stratification by echocardiography and Troponin T in patients with suspected acute coronary syndrome, compared with conventional in-hospital evaluation.

The trial will be conducted at Sørlandet Hospital, Norway. One acute care ambulance in Agder county will be equipped with a high-end cardiac ultrasound scanner with wireless communication to the cardiac centre/cardiologist, and a point-of-care troponin T quantitative analysis kit Paramedics will be offered a comprehensive hands-on course in cardiac ultrasound image acquisition by an echo-technician and a cardiologist. Similar, a short course will be given in point-of-care troponin analysis.

Imaging quality Communication between paramedic and cardiologist established Image transfer and interpretation by cardiologist functional Technical problems addressed and solved in collaboration with manufacturer

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the medical dispatch center (AMK) with chest pain; Norwegian medical index criteria A10.2- A10.11
* Men and women
* Age ≥ 18
* Informed consent for participation
* Examined by paramedics in a prehospital setting due to newly onset (<12 hours) chest pain (lasting for >20 min) and suspected AMI

Exclusion Criteria:

* Any condition which interfere with the ability to cooperate
* Hemodynamic instability
* Severe mental disorder
* Pregnancy or breast-feeding
* STEMI
* Obvious non-cardiac origin of the chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Prehospital identification of Acute coronary syndromes | 1 year
  Evaluate the feasibility of paramedics performing POC Hs-cTnT measurements and focused TTE for prehospital NSTE-ACS risk stratification. Investigate if focused prehospital transthoracic echocardiography (TTE) images achieved by paramedics could be transferred to the in-hospital cardiologist for diagnostic evaluation, and test if this, in combination with a point-of-care (POC) high-sensitive Troponin-T (Hs-cTnT ) test, facilitates prehospital identification of high risk NSTE-ACS. Measure: number of prehospital NSTEMI discovered or missed on the prehospital evaluation, through patient journal review at day 30. and 90.
Transferability of images and test results | 1 year
  Measure if focused prehospital transthoracic echocardiography (TTE) images achieved by paramedics could be transferred to the in-hospital cardiologist for diagnostic evaluation in combination with a point-of-care (POC) high-sensitive Troponin-T (Hs-cTnT ) test. Measure: Quality assessment on 1-5 scale. count of interpretable images.

CONTACTS AND LOCATIONS:
Overall Officials: Jarle Jortveit, PhD HOD, Principal Investigator — Sorlandet Hospital Thrust and Air Ambulance foundation
Locations (1):
- SSHF, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: Yes
Will share anonymized images upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol now accessable on Recearchgate
Access Criteria: Asking Primary investigator for permit
URL: https://www.researchgate.net/

REFERENCES:
- [Derived] Jacobsen L, Grenne B, Olsen RB, Jortveit J. Feasibility of prehospital identification of non-ST-elevation myocardial infarction by ECG, troponin and echocardiography. Emerg Med J. 2022 Sep;39(9):679-684. doi: 10.1136/emermed-2021-211179. Epub 2022 Jan 21. PMID 35064012

DOCUMENTS (1):
  • Study Protocol (2019-12-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT04223986/Prot_000.pdf